CLINICAL TRIAL: NCT06090825
Title: Real World Status of Palliative Care for Pancreatic Cancer Patients in China-a National Multi-center Cross-sectional Survey
Brief Title: Cross-sectional Survey on Palliative Therapy for Pancreatic Cancer Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiaofei Liu, Department director assistant, clinical chief professor, Peking Union Medical College Hospital
Other Study IDs: K4602
Record Dates: First submitted 2023-10-03; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer
Keywords: follow up; palliative care; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic cancer patients
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
It is a real-world observational cross-sectional follow-up study on clinical palliative care for pancreatic cancer patients in China. It is evaluated by an online questionnaire sent to the doctors from the General Surgery Department in more than 100 public tertiary teaching hospitals and about 350 public primary care units in the Chinese mainland.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly malignant gastrointestinal tumor with only a 10% overall 5-year survival rate. More than 80% of patients are already in the advanced stage when diagnosed, losing the chance of surgery. Advanced pancreatic cancer progresses rapidly and chemoradiotherapy has limited efficacy, so palliative care is thought to play an important role in the treatment process. However, due to the late development of palliative care, there is a lack of data on real-world clinical palliative care for pancreatic cancer patients in China.

This study investigates the real-world current status of palliative care for pancreatic cancer patients by sending a web questionnaire to the doctors from the Department of General Surgery in more than 100 public tertiary teaching hospitals and about 350 public primary care units in the Chinese mainland. The survey aims to obtain the real status of palliative care and achieve a comprehensive understanding of how to develop palliative care in hospitals.

The questionnaire includes both subjective standards like the surgeons' opinion on the development of palliative therapy and objective standards such as dedicated beds and teams for palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Doctors from the General Surgery Department in Chinese public tertiary teaching hospitals and public primary care units
* Approval to participate
* Participants with a valid and complete questionnaire evaluated by 2 experienced surgeons

Exclusion Criteria:

* Refusal to participate
* Participants with an invalid or incomplete questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The doctors of the Department of General Surgery in more than 100 public tertiary teaching hospitals and about 350 public primary care units in the Chinese mainland
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Descriptions and scores of real status of hospice care in different hospitals | 1 month
  The primary outcome is objective standards and subjective scores of current status of palliative care to qutify the development of palliative care of different hospitals. The score is evaluated by a follow-up questionnaire. The maximum and minimum score is 10 and 0, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Qiaofei Liu, Study Chair — Department of General Surgery, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No